CLINICAL TRIAL: NCT02744391
Title: A Study of L-DOPA for Depression and Slowing in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7270
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Major Depressive Disorder; Dysthymia; Depression Not Otherwise Specified; Decreased Processing Speed; Decreased Gait Speed
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder | interventions — Levodopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- L-DOPA (Experimental): Patients will receive titration of L-DOPA from 150 mg to 450 mg.
  Interventions: Drug: Levodopa

INTERVENTIONS:
Drug: Levodopa
  Other Names: L-Dopa

SUMMARY:
Individuals with Late Life Depression (LLD) often have cognitive problems, particularly problems with memory, attention, and problem solving, all of which contribute to antidepressant non-response. Our group and others have shown that decreased thinking speed is the central cause of functional problems in patients with LLD. Similarly, decreased walking speed is associated with depression and carries additional risk for falls, hospitalization, and death. Available evidence suggests that declining functionality in the brain's dopamine system contributes to age-related cognitive and motor slowing. The central hypothesis of this R61/R33 Phased Innovation Award is that by enhancing dopamine functioning in the brain and improving cognitive and motor slowing, administration of carbidopa/levodopa (L-DOPA) will improve depressive symptoms in older adults.

DETAILED DESCRIPTION:
This study will elucidate the neurobiology of slowing and LLD, identify a novel therapeutic target for depression, and contribute to the development of personalized treatment regimens for LLD. The multimodal neuroimaging methods detailed in this application will provide information about the neurobiology of aging-associated slowing and LLD at molecular, structural, and functional levels of analysis. These data will fill a crucial gap in our knowledge regarding what are the physiologic and functional consequences of dopamine depletion occurring across the lifespan in individuals without PD. Results from this project also will allow us to evaluate a novel therapeutic approach to LLD, which could have large public health ramifications given the prevalence, frequent treatment resistance, and chronicity characteristic of LLD. Even apart from patients with LLD, cognitive and motor slowing exact a large public health burden in terms of impaired functioning and increased morbidity and mortality, and this burden will only grow as the population ages. It is critical to develop treatments capable of altering the negative health trajectories associated with slowing in order to help older adults maintain independent functioning and live longer with an increased quality of life. Finally, while PET and MRI may prove critical to understand the neurobiology of slowing and LLD, their invasiveness and expense limit their roles in informing treatment decisions in clinical practice settings. For this reason the investigators are also assessing the influence of genetic moderators such as interleukin-6 (IL-6) and catechol-O-methyl-transferase (COMT) genotype on baseline dopamine functioning and response to L-DOPA. This may facilitate the identification of both high-risk individuals and those most likely to benefit from treatment interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age >59 years
* DSM 5 non-psychotic Major Depressive Disorder, Dysthymia, or Depression Not Otherwise Specified
* Center for Epidemiological Studies Depression (CES-D) Rating Scale > 9
* Decreased processing speed (defined as 0.5 SD below age-adjusted norms on the Digit Symbol Test) and decreased gait speed (defined as average walking speed over 15' course < 1 m/s)
* Willing and capable of providing informed consent and complying with study procedures
* Prefer not to be treated with a standard treatment for MDD, Dysthymia, or Depression NOS (e.g., antidepressant medication or psychotherapy)

Exclusion Criteria:

* Diagnosis of substance abuse or dependence (excluding Tobacco Use Disorder) within the past 12 months
* History of or current psychosis, psychotic disorder, mania, or bipolar disorder
* Diagnosis of probable Alzheimer's Disease, Vascular Dementia, or PD
* Mini Mental Status Exam (MMSE) < 25
* HRSD ≥ 25 or the presence of significant suicide risk
* Current or recent (within the past 4 weeks) treatment with antidepressants, antipsychotics, dopaminergic agents, or mood stabilizers
* History of allergy, hypersensitivity reaction, or severe intolerance to LDOPA
* Acute, severe, or unstable medical or neurological illness
* Mobility limiting osteoarthritis of any lower extremity joints, symptomatic lumbar spine disease, history of joint replacement surgery, or history of spine surgery
* Hypotension (SBP<90), hypertension (SBP >150 or DBP > 90), past stroke causing sensory or movement deficits, cardiac arrhythmias, or any other severe or uncontrolled cardiovascular disease
* Having contraindication to MRI scanning (such as metal in body) or unable to tolerate the scanning procedures
* History of significant radioactivity exposure (nuclear medicine studies or occupational exposure)
* Presence of a clinically significant brain abnormality, significant anemia, insulin dependent diabetes, a history of cardiovascular disease, or uncontrolled/untreated risk factors for coronary artery disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained from this study will be shared with the National Institute of Mental Health (NIMH) Data Archive (NDA) and will maintain patient confidentiality by ensuring exclusion of all 18 identifiers (outlined by HIPAA) prior to data sharing. All assessment outcomes will be shared twice a year as per NIMH Data Archive (NDA) guidelines.
Time Frame: Data will be available for as long as NIMH deems necessary.
Access Criteria: Information can be accessed by going to the NUMH Data Archive website and searching the protocol. One must request access to detailed human subjects data. To do this you must be sponsored by an NIH recognized institution with a Federal wide Assurance and have a research related need to access NIMH Data Archive (NDA) data.

REFERENCES:
- [Derived] Wengler K, Ashinoff BK, Pueraro E, Cassidy CM, Horga G, Rutherford BR. Association between neuromelanin-sensitive MRI signal and psychomotor slowing in late-life depression. Neuropsychopharmacology. 2021 Jun;46(7):1233-1239. doi: 10.1038/s41386-020-00860-z. Epub 2020 Sep 12. PMID 32919398
- [Derived] Rutherford BR, Slifstein M, Chen C, Abi-Dargham A, Brown PJ, Wall MW, Vanegas-Arroyave N, Stern Y, Bailey V, Valente E, Roose SP. RETRACTED: Effects of L-DOPA Monotherapy on Psychomotor Speed and [11C]Raclopride Binding in High-Risk Older Adults With Depression. Biol Psychiatry. 2019 Aug 1;86(3):221-229. doi: 10.1016/j.biopsych.2019.04.007. Epub 2019 Apr 15. PMID 31178096

RESULTS

PARTICIPANT FLOW:
Groups:
- L-DOPA: Patients will receive titration of L-DOPA from 150 mg to 450 mg.
  Levodopa
Period: Overall Study
Arm/Group | L-DOPA
Started | 47
Completed | 33
Not Completed | 14
Not completed — Lost to Follow-up | 9
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | L-DOPA
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 26
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47
Hamilton Rating Scale for Depression (24 item) [Mean (Standard Deviation); unit: Units on a scale] — Our target is depressive symptomatology as measured by the Hamilton Rating Scale for Depression (HRSD). The HRSD is a 24-item questionnaire used as an indication of depression and a guide to evaluate recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score of 16 or above is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity. Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
  Units on a scale
    number analyzed (Participants) | 36
    (all) | 15.53 (6.04)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (24 Item)
Description: Our target is depressive symptomatology as measured by the Hamilton Rating Scale for Depression (HRSD). The HRSD is a 24-item questionnaire used as an indication of depression and a guide to evaluate recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score of 16 or above is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity.
Time Frame: Week 3
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
Units on a Scale | 10.94 (6.87)

2. Secondary Outcome: Digit Symbol Substitution Test
Description: Digit symbol substitution test (DSST) is a neuropsychological test sensitive to brain damage, dementia, age and depression. The test is not sensitive to the location of brain-damage (except for damage comprising part of the visual field). It consists of (e.g. nine) digit-symbol pairs (e.g. 1/-,2/┴ ... 7/Λ,8/X,9/=) followed by a list of digits. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time (e.g. 90 or 120 sec) is measured. The higher the number, the better the score.
Time Frame: Screening
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
total score | 31.86 (9.69)

3. Secondary Outcome: Digit Symbol Substitution Test
Description: as for outcome 2
Time Frame: Week 3
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
total score | 41.42 (9.56)

4. Secondary Outcome: Pattern Comparison
Description: This test required participants to identify whether two visual patterns are the "same" or "not the same" (responses were made by pressing a "yes" or "no" button). Patterns were either identical or varied on one of three dimensions: color (all ages), adding/taking something away (all ages), or one versus many. Scores reflected the number of correct items (of a possible 130) completed in 90 s; items were designed to minimize the number of errors that were made.
Time Frame: Screening
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
total score | 24.72 (5.42)

5. Secondary Outcome: Pattern Comparison
Description: as for outcome 4
Time Frame: Week 3
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
total score | 27.61 (4.95)

6. Secondary Outcome: Letter Comparison
Description: Subjects will be asked to determine whether two strings of letters are the same or different. There are 3 pages and the subject is given 30 seconds per page. Scoring is based on the number answered correctly. The higher the number, the better the score.
Time Frame: Screening
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: Total Correct
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
Total Correct | 14.36 (4.73)

7. Secondary Outcome: Letter Comparison
Description: as for outcome 6
Time Frame: Week 3
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: Total Correct
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
Total Correct | 15.69 (4.54)

8. Secondary Outcome: Single Task Gait Speed
Description: Patients' gait will be assessed as walking speed in m/s on a 15' walking course. Patients are instructed to walk at their usual or normal speed for a total of 27' (starting and ending at a point 6 feet prior to and after the 15' course to eliminate acceleration and deceleration effects). Two trials will be completed, and gait speed will be based on the average of 2 trials.
Time Frame: Screening
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
m/s | 0.80 (0.18)

9. Secondary Outcome: Single Task Gait Speed
Description: as for outcome 8
Time Frame: Week 3
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
m/s | .92 (.21)

10. Secondary Outcome: Dual Task Gait Speed
Description: For the Dual Task, patients are instructed to walk at their usual pace while simultaneously verbally listing as many animals as possible. In addition, a counting Dual Task will be used in which patients are instructed to walk at their usual pace while simultaneously performing serial subtractions by three starting at 100. Patients will start and end at a point 2 meters from the Gaitrite mat to eliminate acceleration and deceleration effects. Dual Task will be assessed two times with the average used in the analyses
Time Frame: Screening
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
m/s | 0.69 (.23)

11. Secondary Outcome: Dual Task Gait Speed
Description: For the Dual Task, patients are instructed to walk at their usual pace while simultaneously verbally listing as many animals as possible. In addition, a counting Dual Task will be used in which patients are instructed to walk at their usual pace while simultaneously performing serial subtractions by three starting at 100. Patients will start and end at a point 2 meters from the Gaitrite mat to eliminate acceleration and deceleration effects. Dual Task will be assessed two times with the average used in the analyse.
Time Frame: Week 3
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
m/s | 0.82 (.24)

12. Secondary Outcome: Inventory of Depressive Symptomatology-Self Report
Description: Rating scale for depressive symptoms based on Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria that has been increasingly used in antidepressant studies due to its equivalent weightings for each item, understandable anchor points, and inclusion of all Diagnostic and Statistical Manual of Mental Disorders criteria. Patients will be asked to circle the one response to each item that best describes them for the past seven days. The answers range 0-84. The higher the score the greater the depressive symptoms.
Time Frame: Screening
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
total score | 26.42 (12.57)

13. Secondary Outcome: Inventory of Depressive Symptomatology-Self Report
Description: as for outcome 12
Time Frame: Week 3
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | L-DOPA
Number analyzed (Participants) | 36
total score | 15.09 (10.64)

14. Secondary Outcome: Pre-Treatment [11C]-Raclopride Binding Potential: Sensorimotor Striatum
Description: Subjects received 2 [11C]-raclopride positron emission tomography (PET) scans: baseline and post-L-DOPA treatment. High resolution anatomical T1-weighted MRI scans were acquired for each subject and PET data were co-registered to the MRIs using maximization of mutual information (SPM12, Wellcome Centre for Human Neuroimaging). Regions of interest (ROIs) were applied to the MRIs and transferred to the PET data and included the sensorimotor striatum (post-commissural putamen, SMST), associative striatum (whole caudate and pre-commissural putamen, AST) and the limbic striatum (nucleus accumbens and the most ventral aspects of the pre-commissural caudate and putamen, LST). Additionally, an ROI was drawn on cerebellum as a reference tissue. ROI time activity curves were derived as the average activity in each ROI in each frame. The primary outcome measure was BPND, the binding potential with respect to the non-displaceable compartment, derived by the simplified reference tissue model.
Time Frame: Baseline
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis.
Measure: Mean (Standard Deviation); unit: mCi/ ml
Arm/Group | L-DOPA
Number analyzed (Participants) | 10
mCi/ ml | 2.43 (0.25)

15. Secondary Outcome: Post-Treatment [11C]-Raclopride Binding Potential: Sensorimotor Striatum
Description: as for outcome 14
Time Frame: Week 3
Population: 47 patients were enrolled and 36 patients were analyzed according to the intent to treat analysis. Only 10 subjects were scanned in this study.
Measure: Mean (Standard Deviation); unit: mCi/ ml
Arm/Group | L-DOPA
Number analyzed (Participants) | 10
mCi/ ml | 2.19 (0.29)

16. Secondary Outcome: Pre-Treatment [11C]-Raclopride Binding Potential: Limbic Striatum
Description: as for outcome 14
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mCi/ ml
Arm/Group | L-DOPA
Number analyzed (Participants) | 10
mCi/ ml | 2.04 (0.18)

17. Secondary Outcome: Post-Treatment [11C]-Raclopride Binding Potential: Limbic Striatum
Description: as for outcome 14
Time Frame: Week 3
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mCi/ ml
Arm/Group | L-DOPA
Number analyzed (Participants) | 10
mCi/ ml | 2.04 (0.15)

18. Secondary Outcome: Pre-Treatment [11C]-Raclopride Binding Potential: Associative Striatum
Description: as for outcome 14
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mCi/ ml
Arm/Group | L-DOPA
Number analyzed (Participants) | 10
mCi/ ml | 2.17 (0.26)

19. Secondary Outcome: Post-Treatment [11C]-Raclopride Binding Potential: Associative Striatum
Description: as for outcome 14
Time Frame: Week 3
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mCi/ ml
Arm/Group | L-DOPA
Number analyzed (Participants) | 10
mCi/ ml | 2.05 (0.26)

ADVERSE EVENTS:
Time Frame: 3 Weeks
Arm/Group | L-DOPA
All-Cause Mortality (participants affected / at risk) | 1/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

LIMITATIONS AND CAVEATS:
Data collected in the trial have been presented as required but are considered unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT02744391/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02744391/ICF_001.pdf